CLINICAL TRIAL: NCT06925451
Title: Effects of Natural Sourdough Fermentation Duration and Acid Development on Postprandial Blood Glucose in Prediabetic Adults
Brief Title: Effects of Sourdough Fermentation Duration and Acid Development on Postprandial Blood Glucose in Prediabetic Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Principal Investigator, Carol Johnston, Professor and Senior Associate Dean, Arizona State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: STUDY00021470
Record Dates: First submitted 2025-04-06; First posted 2025-04-13 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-08

CONDITIONS: Insulin Resistance
Keywords: fermentation; pre-diabetes; sourdough bread; post-prandial glycemia
MeSH Terms: conditions — Insulin Resistance; Glucose Intolerance

STUDY DESIGN:
Intervention Model Description: The day prior to testing is standardized: no vigorous activity or alcohol consumption, and two bagels are to be consumed between 3 pm and 8 pm. Participants will begin an overnight fast starting around 10 pm (only water is to be consumed). The bagels will be provided at no charge. For each of the 4 test visits, participants arrive in a fasted state and a blood drop will be collected via finger prick to measure glucose. The 'test meal' will be consumed under observation within 8 minutes. The three fermented versions on the sourdough bread and the control bread will be fed using a four-block randomization process. Finger pricks will take place at 30, 60, 90, and 120 minutes post meal. The participant will be asked to complete hunger measures and report on the acceptability of the bread at the completion of testing.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- sourdough bread 24 (Experimental): 24 hours fermentation
  Interventions: Other: sourdough bread 24
- Control bread (Active Comparator): 12 hours fermentation
  Interventions: Other: yeast bread
- sourdough bread 48 (Experimental): 48 hours fermentation
  Interventions: Other: sourdough bread 48
- sourdough bread 72 (Experimental): 72 hours fermentation
  Interventions: Other: sourdough bread 72

INTERVENTIONS:
Other: sourdough bread 24 — fermentation time=24 hours
  Arms: sourdough bread 24
Other: sourdough bread 48 — fermentation time=48 hours
  Arms: sourdough bread 48
Other: sourdough bread 72 — fermentation time=72 hours
  Arms: sourdough bread 72
Other: yeast bread — no fermentation
  Arms: Control bread

SUMMARY:
The primary intervention for management of prediabetes is lifestyle changes. Eating healthier and increasing physical activity was found to slow the progression of prediabetes into diabetes, reduce the risk of other diseases like cardiovascular disease and hypertension, and have a lasting impact even after the intervention is discontinued. Studies found that increasing the intake of fiber, pre- and probiotics, and fermented foods have been linked to improved glycemic biomarkers. The goal of this crossover randomized trial is to assess the relationship between lengthened fermentation time of sourdough bread, e.g., an increased amount of lactic acid and acetic acid in the bread product, and postprandial glycemic response in healthy adults with prediabetes.

DETAILED DESCRIPTION:
Sourdough bread has been proven to have higher fiber content and contains beneficial microorganisms from the fermentation process and has been linked to reduced risk of various diseases like diabetes, cardiovascular disease, and dyslipidemia. The fermentation of sourdough bread products converts starch and sugar in the dough into resistant starches and other slower digesting compounds. Sourdough bread products also have a lower glycemic index value, meaning they do not cause the blood sugar to rise as quickly, thus slowing the release of insulin in the body, leading to reduced risk of insulin resistance. However, very few studies exist studying the effects of naturally fermented sourdough products in individuals with prediabetes. It is worth exploring if increasing the fermentation time of naturally fermented sourdough bread increases the effects on relevant biomarkers relating to postprandial glycemia and insulinemia in prediabetic adults.

This study examined the acute effect of varying lengths of sourdough fermentation times on postprandial blood glucose levels over a 4-week period in adults with prediabetes (as evidenced by fasting glucose ≥100 or diagnosis by physician), but not taking diabetic medications. For each trial, the sourdough bread was ingested after an overnight fasting period in order to evaluate the effects of the bread when incorporated into the diet in place of breads made with baker's yeast. The goal of this crossover randomized trial was to assess the relationship between lengthened fermentation time, meaning an increased amount of lactic acid and acetic acid in the bread product, and glycemic and insulinemic response.

ELIGIBILITY:
Inclusion Criteria:

* prediabetes; not on metformin; no known food allergies or sensitivities; not supplementing pre/post biotics

Exclusion Criteria:

* following diet that restricts carbohydrates; medication use affecting blood glucose; acute illness; smoker; pregnant; lactating; GI tract surgery; not willing to follow protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2025-04-04 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
blood glucose | conducted at fasting and 30, 60, 90, and 120 minutes post-meal
  blood glucose will be measured using a glucometer and capillary blood from finger prick

SECONDARY OUTCOMES:
hunger rating | conducted at 120 minutes post-meal
  Hunger rating will be determined using Likert scale. Anchors: not hungry at all and as hungry as I have ever felt. A higher score indicates greater hunger.
bread palatability | conducted at 120 minutes post-meal
  bread palatability will be measured by Likert scale

CONTACTS AND LOCATIONS:
Locations (1):
- 850 PBC, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to publish in ICMJE journals